CLINICAL TRIAL: NCT06046092
Title: An Open Label, Dose Escalation Phase I Trial to Assess Safety and Immunogenicity of the H7HLAII DNA Vaccine, Encoding Influenza Hemagglutinin H7 Directed to HLA Class II, for Prophylaxis of Pandemic Influenza Infection in Healthy Volunteers
Brief Title: H7HLAII DNA Influenza Vaccine
Acronym: H7N9vax-1
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Gunnveig Grødeland, Coordinating Investigator, Oslo University Hospital
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 2022-500706-18-01
Record Dates: First submitted 2023-09-03; First posted 2023-09-21 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Influenza A; Pandemic Influenza

STUDY DESIGN:
Intervention Model Description: Open label, single arm dose escalation phase I trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Vaccinated (Experimental): Participants will be allocated to one of 3 dose groups, each receiving two intradermal (i.d.) vaccinations with 0.12 mg, 0.60 mg, or 3.00 mg of H7HLAII, respectively.
  Interventions: Biological: H7HLAII

INTERVENTIONS:
Biological: H7HLAII — DNA vaccine encoding influenza hemagglutinin (HA) from influenza A/Shanghai/2/2013 (H7N9) directed to cells expressing human leukocyte antigen class II (HLAII) molecules

SUMMARY:
The purpose of this study is to assess safety and immunogenicity of H7HLAII, a DNA vaccine encoding influenza hemagglutinin (HA) from influenza A/Shanghai/2/2013 (H7N9) directed to cells expressing human leukocyte antigen class II (HLAII) molecules, for prophylaxis of pandemic H7N9 influenza infection in healthy volunteers.

DETAILED DESCRIPTION:
H7HLAII is a DNA vaccine that could remedy the current challenges of slow production for conventional influenza vaccines. The prolonged production time of current influenza vaccines has as a consequence that circulating influenza strains often have drifted significantly from the vaccine included strains, and as such reducing vaccine efficacy. The rapid production enabled by the DNA format could enhance efficacy of seasonal influenza vaccines, but is particularly well suited for prophylaxis against an emerging influenza pandemic.

The only vaccine format that can presently be produced and deployed within 2-3 months is DNA. However, DNA vaccines are typically hampered by low immunogenicity. To surpass this challenge, H7HLAII genetically links the influenza H7 HA to a targeting unit that steers the produced vaccine proteins to HLA class II expressing antigen presenting cells (APC). Previously, this strategy has been shown to increase immunogenicity after vaccination in mice, ferrets, pigs, and rhesus macaques, with a particular strength in antibody induction. Of note, antibodies represent a correlate of protection against influenza, as well as most other infectious diseases. It has also been shown that H7HLAII protected immunized ferrets against a homologous H7N9 strain, and with no safety concerns after toxicity testing in guinea pigs.

H7HLAII is designed to induce strong antibody responses against a specific strain of H7N9 influenza. At present, there are several strains of H7N9 that cause concern for future pandemic emergences, in that periodic zoonotic transmissions are observed in Asia. To date, H7N9 viruses do not have the ability to transmit between humans, but the high mortality rates observed after zoonotic transmissions dictates that society ought to be ready for future emergences. H7HLAII is designed to enable rapid exchange of antigen, allowing for accommodation of any HA into the vaccine construct. As such, the strategy could be of great importance for global prophylactic prevention.

Although a pandemic situation might opt for rapid testing, this trial is planned as a cautious phase I trial with healthy volunteers. It should be noted that the safety aspects for a number of DNA vaccines has been good during clinical testing over the past decade, and the first DNA vaccine was recently licensed for human use.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects, as concluded from the medical history, physical examination test including normal vital signs, and clinical judgment, without the need for medication.
* For women with childbearing potential (WOCBP), defined as fertile following menarche and until becoming post-menopausal (i.e. no menses for 12 months without an alternative medical cause) unless permanently sterile by hysterectomy, bilateral salpingectomy and bilateral oophorectomy: Must use a highly effective contraceptive measures (from 4 weeks prior to the first vaccination until 4 weeks after the second vaccination), and a negative urine pregnancy test before administration of each dose of vaccine. Must agree to not donate eggs during the study and the first three months after their last study visit.
* Able to understand and willing to sign the Informed Consent Form (ICF), which includes compliance with the requirements and restrictions listed in the ICF and in this protocol.
* Subjects able to understand and comply with the study protocol, including being able to attend the scheduled visits.

Exclusion Criteria:

* Medical Conditions

  1. Ongoing or recent (< 2 weeks) intercurrent febrile condition
  2. Previous reports of autoimmune disease
  3. Concurrent chronic active viral hepatitis B or C or HIV
  4. BMI>30
  5. Persons with a history of anaphylaxis or serious reactions to a prior vaccination
  6. Persons with known hypersensitivity to any of the vaccine components
  7. Persons who have had a temperature >38 °C during the previous 72 hours
  8. Persons who have had an acute respiratory infection during the last 7 days
  9. Persons who have abnormal electrocardiogram (ECG)
  10. Women who are pregnant or breast-feeding (women of child-bearing potential must have a negative pregnancy test at screening)
  11. Have received any vaccination within the last month
* Prior/Concomitant Therapy 12. Currently taking anti-inflammatory or immunosuppressive drugs 13. Currently taking antibiotics, steroids, phenytoin, chemotherapy, or other immunosuppressive drugs
* Prior/Concurrent Clinical Study Experience 14. Persons who have participated in another clinical trial during the last month
* Diagnostic assessments 15. Abnormal values of the hematologic and clinical chemistry parameters, as judged by the Investigator, including creatinine, AST, ALT (SGPT), bilirubin and alkaline phosphatase values above normal reference values 16. Positive autoantibodies (anti-nuclear antigens, rheumatoid factor) 17. Serum IgG and IgM lower or higher than the normal reference levels 18. Positive serology tests for hepatitis B or C with detectable hepatitis B HBsAg or DNA, or hepatitis C RNA 19. Positive HIV serology test

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Estimated)
Dates: Start 2023-07-15 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Solicited adverse events following vaccination | 10 days
  Solicited injection site reactions: Redness, Swelling, Pain, Erythema, and Induration; Solicited systemic reactions: Fever, Sweating, Chill, Nausea, Diarrhea, Headache, Fatigue, Myalgia, Arthralgia, and Respiratory symptoms.
Abnormalities in physical examination, vital signs, and clinical laboratory tests | 6 months
  Number of participants with aberrant results.

SECONDARY OUTCOMES:
Changes in virus neutralization assay titres relative to baseline | 6 months
  geometric mean titres
Changes in anti-H7 antibody levels relative to baseline | 6 months
  seroconversion rates

CONTACTS AND LOCATIONS:
Overall Officials: Dag Kvale, MSc/PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grodeland G, Fredriksen AB, Loset GA, Vikse E, Fugger L, Bogen B. Antigen Targeting to Human HLA Class II Molecules Increases Efficacy of DNA Vaccination. J Immunol. 2016 Nov 1;197(9):3575-3585. doi: 10.4049/jimmunol.1600893. Epub 2016 Sep 26. PMID 27671110